CLINICAL TRIAL: NCT04150705
Title: A Pilot Study of PET/MR for Rectal Cancer Treatment Monitoring and Surveillance
Brief Title: PET/MR for Rectal Cancer Treatment Monitoring and Surveillance
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: It was determined that the trial could stop early due to surpassing the feasibility rate.
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 201908228
Record Dates: First submitted 2019-10-31; First posted 2019-11-05 (Actual); Results first posted 2023-02-13 (Actual); Last update posted 2023-02-14 (Actual); Status verified 2023-02

CONDITIONS: Rectal Cancer; Cancer of the Rectum
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- FDG PET/MRI (Experimental): -Patients will undergo FDG-PET/MRI in lieu of the standard pelvic MRI at up to 6 time-points at which it would normally be performed in their care for the period of time extending 30-36 months from the time of enrollment (depending on enrollment point). In the surveillance period, when patients typically undergo pelvic MRI every 3 months, the FDG-PET/MRI will be done in lieu of the standard pelvic MRI on an approximately every-other-scan basis. In other words, the FDG-PET/MRI will occur roughly once every 6 months.
  Interventions: Device: FDG PET/MRI

INTERVENTIONS:
Device: FDG PET/MRI — -All patients will undergo a simultaneous list mode PET and MR acquisition beginning 55-65 minutes after administration of FDG according to a standard weight-based scale.

SUMMARY:
The goal of pilot study is to assess the feasibility of FDG-PET/MRI for monitoring rectal cancer disease status in the setting of rectal cancer non-operative management (NOM). Data from this study will be used to guide the design of future clinical trials involving FDG-PET/MRI for rectal cancer NOM.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age
* Biopsy-proven rectal adenocarcinoma of the rectum with clinically suspected or previously known stage I-IIIB (cT1-4, N0-2, M0) disease
* Anticipated or prior chemoradiation as part of an NOM treatment strategy
* Ability to understand and willingness to sign an IRB-approved written informed consent document

Exclusion Criteria:

* Prior surgical resection of rectal cancer (endoscopic or TME)
* Contraindication to MRI
* Comorbidities that would limit patient's ability to cooperate with a PET/MRI examination (e.g. dementia, inability to follow commands, claustrophobia, tremors, requirement for oxygen by nasal cannula, etc…).
* Implanted devices or materials that may interfere with MRI imaging or create significant artifact
* Pregnancy
* Contraindication to gadolinium contrast or FDG
* End-stage renal disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2022-09-01 (Actual); Study Completion 2022-09-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tyler Fraum, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | FDG PET/MRI
Started | 14
Completed | 14
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | FDG PET/MRI
Number analyzed (Participants) | 14
Age, Continuous [Median (Full Range); unit: years] | 51.6 [38.4 to 83.3]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 14
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 13
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 14

OUTCOME MEASURES:

1. Primary Outcome: Technical Feasibility of PET/MRI as Measured by the Completion of the Study With Acceptable Image Quality in ≥70% of Scans
Description: -For patients imaged at multiple time points after enrollment, all available PET/MRIs will be included in the feasibility analysis. Patients able to remain on the scanner for the full duration of the planned data acquisition without any serious adverse events will be considered to have completed the PET/MRI rectal cancer protocol. Image quality will be assessed by the Principal Investigator on review at a dedicated workstation with specialized PET/MR software. A standardized Likert-based scoring scheme will be utilized to capture subjective assessments of image contrast (1 = worst; 5 = best), image resolution (1 = worst; 5 = best), and image artifact 'freeness' (1 = worst; 5 = best). Image sets scoring ≥ 3 in all three categories will be considered of acceptable quality.
Time Frame: Up to 12 months after completion of enrollment of all patients (26 months)
Measure: Number; unit: percentage of scans that were acceptable
Units Other Than Participants: PET/MRI scans
Arm/Group | FDG PET/MRI
Number analyzed (Participants) | 14
Number analyzed (PET/MRI scans) | 23
percentage of scans that were acceptable | 95.65

2. Secondary Outcome: Percentage of Scans With Changes in Perceived Disease Status as Measured by PET/MRI Tumor Regression Grade Relative to the Conventional MRI Only Tumor Regression Grade
Description: * The study reader will interpret the MRI for the tumor regression grade and then will interpret the PET/MRI for the tumor regression grade.
  * The tumor regression grade is a five-tier imaging-based scoring system based on the ability to distinguish between tumor and fibrosis. mrTRG 1, low signal fibrosis only, no tumor signal; mrTRG 2, more than 75 per cent fibrosis and minimal tumor signal intensity; mrTRG 3, 50 per cent tumor/fibrosis; mrTRG 4, less than 25 per cent fibrosis, predominant tumor signal; and mrTRG 5, no fibrosis
Time Frame: Up to 12 months after completion of enrollment of all patients (26 months)
Population: 7 participants were evaluable for this outcome measure as they were deemed to not be immediate surgical candidates and went on to receive total neoadjuvant therapy (TNT).
Measure: Number; unit: percentage of scans
Units Other Than Participants: PET/MRI scans
Arm/Group | FDG PET/MRI
Number analyzed (Participants) | 7
Number analyzed (PET/MRI scans) | 11
percentage of scans | 18.18

ADVERSE EVENTS:
Time Frame: Adverse events were collected for a period of 24 hours following the administration of the radiotracer FDG.
Arm/Group | FDG PET/MRI
All-Cause Mortality (participants affected / at risk) | 0/14
Serious Adverse Events (participants affected / at risk) | 0/14
Other Adverse Events (participants affected / at risk) | 2/14
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | FDG PET/MRI (N=14)
Nausea (Gastrointestinal disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-07-14): https://cdn.clinicaltrials.gov/large-docs/05/NCT04150705/Prot_SAP_000.pdf